CLINICAL TRIAL: NCT03571659
Title: To Assess the Safety and Efficacy of Two Subthreshold Parameters (5% and 15% Duty Cycle (DC)) Compared to Standard ETDRS (Early Treatment of Diabetic Retinopathy Study) Continuous Wave (CW) Laser
Brief Title: Comparison of Different Fluence Settings for Yellow Subthreshold Laser Treatment in Diabetic Macular Edema
Status: Completed | Type: Observational
Sponsor: L.V. Prasad Eye Institute (Other)
Responsible Party: Principal Investigator, Dr Jay Chhablani, Principal Investigator, L.V. Prasad Eye Institute
Other Study IDs: LVPEI-2018
Record Dates: First submitted 2018-05-18; First posted 2018-06-27 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Lasers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- two subthreshold parameters: 5% and 15% duty cycle (DC)
  Interventions: Procedure: Laser
- standard ETDRS: early treatment of diabetic retinopathy study
  Interventions: Procedure: Laser

INTERVENTIONS:
Procedure: Laser

SUMMARY:
To assess the safety and efficacy of two subthreshold parameters (5% and 15% duty cycle (DC)) compared to standard ETDRS (early treatment of diabetic retinopathy study) continuous wave (CW) laser

DETAILED DESCRIPTION:
Test burn up to barely visible burn with micropulse laser, then reduce the power by 70% and perform laser with various DC (5%, 15%, cw) as per the group.

Focal to Mas+ confluent burns to areas of diffuse leakage

ELIGIBILITY:
Inclusion Criteria:

* Eyes with DME (center or non-center involving) with <350 microns central retinal thickness

Exclusion Criteria:

* Subfoveal exudates, history of VR surgery, history of macular laser

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asian
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2014-12-22 (Actual); Primary Completion 2014-12-22 (Actual); Study Completion 2015-08-11 (Actual)

PRIMARY OUTCOMES:
1. Decrease in number of leaking Mas on FFA 2. Decrease in diffuse leakage on FFA | 3 months
  Comparing the number of leaking microaneuyrms baseline to 6 weeks with 3 types of lasers (two subthreshold parameters (5% and 15% duty cycle (DC)) compared to standard ETDRS continuous wave (CW) laser.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chhablani J, Alshareef R, Kim DT, Narayanan R, Goud A, Mathai A. Comparison of different settings for yellow subthreshold laser treatment in diabetic macular edema. BMC Ophthalmol. 2018 Jul 11;18(1):168. doi: 10.1186/s12886-018-0841-z. PMID 29996798